CLINICAL TRIAL: NCT04975425
Title: Effects of Guiding Catheter on Fractional Flow Reserve and Non-Hyperemic Pressure Ratios for the Assessment of Coronary Artery Stenoses - Disengage @Rest
Brief Title: Effects of Guiding Catheter on FFR and NHPR for the Assessment of Coronary Artery Stenoses (Disengage@Rest)
Acronym: Disengage@Rest
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, Full Professor of Cardiology, Federico II University
Other Study IDs: 3221
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
Keywords: Fractional Flow Reserve; Resting Full-Cycle Ratio
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional Flow Reserve — Comparison between FFR and NHPR before and after guiding catheter disengagement
  Other Names: RFR; Pd/Pa

SUMMARY:
The DISENGAGE@rest study is a prospective registry carried out at Federico II University of Naples with the aim to evaluate the influence of the guiding catheter engagement within the coronary ostium on both FFR and non-hyperaemic pressure ratios values (such as Pd/Pa and the Resting Full-cycle Ratio -RFR), as well as the corresponding clinical impact on decision-making strategies. Consecutive patients with at least one intermediate stenosis (40%-90% by visual estimation) in any of the 3 main coronary arteries will be included.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients provides informed consent;
* Documented coronary artery disease:
* chronic coronary syndromes
* acute coronary syndromes presenting with at least one stenosis with indication for invasive functional assessment.

Exclusion Criteria:

* Patients unable to provide informed consent;
* Pregnant women;
* Any contraindication to perform angiographic study or functional evaluation with pressure wire;
* Patients with aorto-ostial stenosis
* Target vessel diameter < 2mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient > 18 years old with coronary artery disease and indication to perform functional assessment
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Differences between FFR before and after guiding catheter disengagement | 10 minutes
  Evaluate the influence of the guiding catheter engagement within the coronary ostium on FFR values.
1. Differences between NHPR before and after guiding catheter disengagement | 10 minutes
  Evaluate the influence of the guiding catheter engagement within the coronary ostium on NHPR values

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben Ahmed H, Bouzouita K, Hamdi I, Boussaid H, Mokaddem A, Ben Ameur Y, Boujnah MR. [Limits of quantitative coronary angiography (QCA) in intermediate stenosis measuring: a correlation and concordance study with intravascular ultrasound (IVUS)]. Tunis Med. 2014 Jun;92(6):373-8. French. PMID 25741837
- [Background] Johnson NP, Toth GG, Lai D, Zhu H, Acar G, Agostoni P, Appelman Y, Arslan F, Barbato E, Chen SL, Di Serafino L, Dominguez-Franco AJ, Dupouy P, Esen AM, Esen OB, Hamilos M, Iwasaki K, Jensen LO, Jimenez-Navarro MF, Katritsis DG, Kocaman SA, Koo BK, Lopez-Palop R, Lorin JD, Miller LH, Muller O, Nam CW, Oud N, Puymirat E, Rieber J, Rioufol G, Rodes-Cabau J, Sedlis SP, Takeishi Y, Tonino PA, Van Belle E, Verna E, Werner GS, Fearon WF, Pijls NH, De Bruyne B, Gould KL. Prognostic value of fractional flow reserve: linking physiologic severity to clinical outcomes. J Am Coll Cardiol. 2014 Oct 21;64(16):1641-54. doi: 10.1016/j.jacc.2014.07.973. PMID 25323250
- [Background] Toth G, Hamilos M, Pyxaras S, Mangiacapra F, Nelis O, De Vroey F, Di Serafino L, Muller O, Van Mieghem C, Wyffels E, Heyndrickx GR, Bartunek J, Vanderheyden M, Barbato E, Wijns W, De Bruyne B. Evolving concepts of angiogram: fractional flow reserve discordances in 4000 coronary stenoses. Eur Heart J. 2014 Oct 21;35(40):2831-8. doi: 10.1093/eurheartj/ehu094. Epub 2014 Mar 18. PMID 24644308
- [Background] Adjedj J, De Bruyne B, Flore V, Di Gioia G, Ferrara A, Pellicano M, Toth GG, Bartunek J, Vanderheyden M, Heyndrickx GR, Wijns W, Barbato E. Significance of Intermediate Values of Fractional Flow Reserve in Patients With Coronary Artery Disease. Circulation. 2016 Feb 2;133(5):502-8. doi: 10.1161/CIRCULATIONAHA.115.018747. Epub 2016 Jan 5. PMID 26733607
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] De Bruyne B, Fearon WF, Pijls NH, Barbato E, Tonino P, Piroth Z, Jagic N, Mobius-Winckler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd K, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Limacher A, Nuesch E, Juni P; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI for stable coronary artery disease. N Engl J Med. 2014 Sep 25;371(13):1208-17. doi: 10.1056/NEJMoa1408758. Epub 2014 Sep 1. PMID 25176289
- [Background] Adjedj J, Toth GG, Johnson NP, Pellicano M, Ferrara A, Flore V, Di Gioia G, Barbato E, Muller O, De Bruyne B. Intracoronary Adenosine: Dose-Response Relationship With Hyperemia. JACC Cardiovasc Interv. 2015 Sep;8(11):1422-1430. doi: 10.1016/j.jcin.2015.04.028. PMID 26404193
- [Background] Gruntzig AR, Senning A, Siegenthaler WE. Nonoperative dilatation of coronary-artery stenosis: percutaneous transluminal coronary angioplasty. N Engl J Med. 1979 Jul 12;301(2):61-8. doi: 10.1056/NEJM197907123010201. PMID 449946
- [Background] van de Hoef TP, Lee JM, Echavarria-Pinto M, Koo BK, Matsuo H, Patel MR, Davies JE, Escaned J, Piek JJ. Non-hyperaemic coronary pressure measurements to guide coronary interventions. Nat Rev Cardiol. 2020 Oct;17(10):629-640. doi: 10.1038/s41569-020-0374-z. Epub 2020 May 14. PMID 32409779
- [Background] Jeremias A, Maehara A, Genereux P, Asrress KN, Berry C, De Bruyne B, Davies JE, Escaned J, Fearon WF, Gould KL, Johnson NP, Kirtane AJ, Koo BK, Marques KM, Nijjer S, Oldroyd KG, Petraco R, Piek JJ, Pijls NH, Redwood S, Siebes M, Spaan JAE, van 't Veer M, Mintz GS, Stone GW. Multicenter core laboratory comparison of the instantaneous wave-free ratio and resting Pd/Pa with fractional flow reserve: the RESOLVE study. J Am Coll Cardiol. 2014 Apr 8;63(13):1253-1261. doi: 10.1016/j.jacc.2013.09.060. Epub 2013 Nov 6. PMID 24211503
- [Background] Svanerud J, Ahn JM, Jeremias A, van 't Veer M, Gore A, Maehara A, Crowley A, Pijls NHJ, De Bruyne B, Johnson NP, Hennigan B, Watkins S, Berry C, Oldroyd KG, Park SJ, Ali ZA. Validation of a novel non-hyperaemic index of coronary artery stenosis severity: the Resting Full-cycle Ratio (VALIDATE RFR) study. EuroIntervention. 2018 Sep 20;14(7):806-814. doi: 10.4244/EIJ-D-18-00342. PMID 29790478
- [Background] Mamas MA, Horner S, Welch E, Ashworth A, Millington S, Fraser D, Fath-Ordoubadi F, Neyses L, El-Omar M. Resting Pd/Pa measured with intracoronary pressure wire strongly predicts fractional flow reserve. J Invasive Cardiol. 2010 Jun;22(6):260-5. PMID 20516504
- [Background] van Nunen LX, Zimmermann FM, Tonino PA, Barbato E, Baumbach A, Engstrom T, Klauss V, MacCarthy PA, Manoharan G, Oldroyd KG, Ver Lee PN, Van't Veer M, Fearon WF, De Bruyne B, Pijls NH; FAME Study Investigators. Fractional flow reserve versus angiography for guidance of PCI in patients with multivessel coronary artery disease (FAME): 5-year follow-up of a randomised controlled trial. Lancet. 2015 Nov 7;386(10006):1853-60. doi: 10.1016/S0140-6736(15)00057-4. Epub 2015 Aug 30. PMID 26333474
- [Background] Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, Engstrom T, Kaab S, Dambrink JH, Rioufol G, Toth GG, Piroth Z, Witt N, Frobert O, Kala P, Linke A, Jagic N, Mates M, Mavromatis K, Samady H, Irimpen A, Oldroyd K, Campo G, Rothenbuhler M, Juni P, De Bruyne B; FAME 2 Investigators. Five-Year Outcomes with PCI Guided by Fractional Flow Reserve. N Engl J Med. 2018 Jul 19;379(3):250-259. doi: 10.1056/NEJMoa1803538. Epub 2018 May 22. PMID 29785878
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Toth GG, Johnson NP, Jeremias A, Pellicano M, Vranckx P, Fearon WF, Barbato E, Kern MJ, Pijls NH, De Bruyne B. Standardization of Fractional Flow Reserve Measurements. J Am Coll Cardiol. 2016 Aug 16;68(7):742-53. doi: 10.1016/j.jacc.2016.05.067. PMID 27515335
- [Background] Pellicano M, Ciccarelli G, Xaplanteris P, Di Gioia G, Milkas A, Colaiori I, Heyse A, Van Durme F, Vanderheyden M, Bartunek J, De Bruyne B, Barbato E. DISENGAGE Registry. Circ Cardiovasc Interv. 2020 Nov;13(11):e008640. doi: 10.1161/CIRCINTERVENTIONS.119.008640. Epub 2020 Nov 2. PMID 33131299